CLINICAL TRIAL: NCT06496659
Title: Segmentectomy After Induction Therapy (SAINT): Phase II Single Arm Trial Evaluating Segmentectomy in Accomplishing R0 Resection for Patients with Lung Cancer Treated with Neoadjuvant Therapy
Brief Title: Segmentectomy After Induction Therapy (SAINT)
Acronym: SAINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Comprehensive Cancer Center of Northwestern University (Unknown)
Responsible Party: Principal Investigator, Ankit Bharat, Chief of Thoracic Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00219945; NU 23L02 (Other: Robert H. Lurie Comprehensive Cancer Center of Northwestern University)
Record Dates: First submitted 2024-05-14; First posted 2024-07-11 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Segmentectomy
Keywords: Non-Small Cell Lung Cancer; Neoadjuvant therapy; Anatomic resection; Post-induction therapy; Surgical intervention
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Segmentectomy after Induction Therapy (Other): Surgical intervention (segmentectomy) post induction therapy for Non-Small Cell Lung Cancer
  Interventions: Procedure: Segmentectomy

INTERVENTIONS:
Procedure: Segmentectomy — A segmentectomy is a surgical procedure to remove a segment of the lung. This surgery will be done on patients who have completed neoadjuvant therapy for diagnosis of Non-Small Cell Lung Cancer.

SUMMARY:
The primary objective will be to determine the feasibility of performing a high-quality sublobar anatomic resection (segmentectomy) with R0 margin status on final pathology for patients who received induction therapy for NSCLC and are downstaged to ≤ycT1cN0M0 (TDi 3cm or less). T1c is tumor staging 1 and c stands for tumor is considered larger than 2cm but no larger than 3cm across; N0 is No regional lymph node metastasis; M0 is No distant metastasis.

DETAILED DESCRIPTION:
With the advent of effective neoadjuvant therapies, many patients with Stage II or III lung cancer are being downstaged to Stage I. Recent studies have shown that sublobar resections, especially segmentectomy, offer superior long-term survival and quality of life for patients with Stage I cancer. However, aside from isolated cases, the safety and feasibility of performing segmentectomy on patients who were initially diagnosed with advanced-stage cancer but were later downstaged to Stage I remain unexplored. Thus, our hypothesis is that segmentectomy can be safely executed in these downstaged Stage I patients after neoadjuvant therapy, without necessitating a conversion to lobectomy due to technical complications. Both segmentectomy and lobectomy are considered standard-of-care lung resection procedures.

Recent randomized clinical trials have demonstrated high rates of pathological downstaging for locally advanced lung cancer treated with neoadjuvant chemoimmunotherapy with R0 resection rates of 83.2% to 77.8% in recent historical controls. Other recent trials demonstrated that high-quality segmentectomy is associated with improved overall survival and is now standard-of-care for early-stage lung cancer with small tumor sizes. Given these findings, the logical next step is to determine if the benefits of high-quality segmentectomy may be extended to an increasingly common clinical scenario where locally advanced lung cancers are downstaged to small tumor size after induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed non-small-cell lung cancer that is clinically staged as ≤ycT1cN0M0 (tumor size 3cm or less on greatest dimension measured by cross-sectional imaging) after receiving induction therapy.
* Patients may have received any regimen of neoadjuvant chemotherapy, neoadjuvant immunotherapy, or neoadjuvant chemoimmunotherapy.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.
* Patients must be age ≥ 18 years.
* Patients must exhibit a/an ECOG (Eastern Cooperative Oncology Group) performance status of <3.
* Patients must have adequate organ function as defined below: These are guidelines that may or should be modified based on protocol-specific or drug development-specific needs.

Table 1: Measures of Adequate Organ Function. FEV1 or DLCO ≥40% (DLCO: diffusing capacity of lung for carbon monoxide)

* For patients with a known history of Human immunodeficiency virus (HIV), infected patients on effective anti-retroviral therapy must have a viral load undetectable for 6 months prior to registration.
* For patients with a known history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be considered a candidate for surgical resection under general anesthesia.
* Females of child-bearing potential (FOCBP) must have a negative pregnancy test prior to registration on study.

NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy
* Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)

Exclusion Criteria:

* Patients who have had prior lung resection or thoracic surgery.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Patients who are receiving any other investigational agents.
* Patients with evidence of distant metastases including brain metastases will be excluded from this study because they will not benefit from surgical resection.
* Patients that do not have documented consensus agreement on the feasibility of anatomic sublobar resection (segmentectomy) from at least 2 study surgeons will not be enrolled.
* Patients with pre-induction therapy tumor involving greater than 1 lobe.
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Hypertension that is not controlled on medication
  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant. Pregnant patients are excluded from this study because the study protocol requires frequent cross-sectional imaging with potential for teratogenic effects.
* Patients with another malignancy within 3 years (except for non-melanoma skin cancer, CIS of cervix (a preinvasive carcinomatous change of the cervix), superficial bladder cancer). Patients with prior malignancies are excluded to isolate overall survival outcomes.
* Patients with active smoking status or cessation <4 weeks prior to surgical resection.
* Patients with biopsy positive hilar or mediastinal lymph nodes following induction therapy detected by EBUS (endobronchial ultrasound), mediastinoscopy, or intraoperative sampling.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2029-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Segmentectomy and R0 on final pathology | Up to 48 hours after date of surgical resection
  The primary objective will be to determine the feasibility of performing a high-quality sublobar anatomic resection (segmentectomy) with R0 margin status on final pathology for patients who received induction therapy for NSCLC and are downstaged to ≤ycT1cN0M0 (TDi 3cm or less).
  To address the primary objective, the proportion of patients who receive high-quality segmentectomy will be determined immediately at the end of the operation and R0 rates on final pathology will be collected after the surgical operation when pathological reports are completed.

SECONDARY OUTCOMES:
R0 resection rates - on final pathology (post-surgery) if converted to lobectomy | Up to 48 hours after date of surgical resection
  The proportion of patients who received lobectomy with R0 resection on final pathology (post-surgery).
Ability to complete the intended procedure (sublobar anatomic resection) | Up to 24 hours after date of surgical resection
  The proportion of patients with completion of the intended procedure (sublobar anatomic resection) based on the extent of surgical resection immediately at the end of the operation
Conversion to lobectomy in a separate operation from sublobar anatomic resection | Up to 6 weeks after date of surgical resection
  The proportion of patients who were converted to lobectomy during the operation or within six weeks after the operation for patients who undergo revision.
Safety, measured as perioperative outcomes (Post-operative length of stay) | Up to 30 days after date of surgical resection
  Safety, measured as perioperative outcomes for patients who receive lobectomy or sublobar anatomic resection (post-operative length-of-stay):
  • Post-operative length of stay defined from the date of surgery until hospital discharge.
  -Outcome measured in number of days
Safety, measured as perioperative outcomes (post-operative discharge destination) | Up to 30 days after date of surgical resection
  Safety, measured as perioperative outcomes for patients who receive lobectomy or sublobar anatomic resection (post-operative discharge destination)
  • Post-operative discharge destination defined as including: i. Home ii. Extended Care/ Transitional Care Unit/ Rehab iii. Other Hospital iv. Nursing Home v. Hospice vi. Other vii. Expired
Safety, measured as perioperative outcomes (time to chest tube removal) | Up to 30 days after date of surgical resection
  Safety, measured as perioperative outcomes for patients who receive lobectomy or sublobar anatomic resection (time to chest tube removal)
  -Outcome measured as number of days from date of surgical resection to time of chest tube removal
Safety, measured as perioperative outcomes (blood transfusion requirements) | Up to 30 days after date of surgical resection
  Safety, measured as perioperative outcomes for patients who receive lobectomy or sublobar anatomic resection (blood transfusion requirements)
  -Outcome measured as number of units blood transfused, if required
Safety, measured as perioperative outcomes (30-day unplanned readmission) | Up to 30 days after date of surgical resection
  Safety, measured as perioperative outcomes for patients who receive lobectomy or sublobar anatomic resection (30-day unplanned readmission)
  -Outcome measured as number of days if unplanned readmission required after date of discharge following surgical resection and reasoning for readmission
Safety, measured as perioperative outcomes (30-day morbidity) | Up to 30 days after date of surgical resection
  Safety, measured as perioperative outcomes for patients who receive lobectomy or sublobar anatomic resection (30-day morbidity)
  -Outcome measured as status of participant at 30 days post-discharge from surgical resection procedure (alive or deceased)
Safety, measured as perioperative outcomes (30-day mortality) | Up to 30 days after date of surgical resection
  Safety, measured as perioperative outcomes for patients who receive lobectomy or sublobar anatomic resection (30-day mortality)
  -Outcome measured as date of death within 30 days following discharge from surgical resection procedure
Change in pre-operative FEV1 (forced expiratory volume at one second) at 3 and 6 months for lobectomy and sublobar anatomic resection | Prior to surgical resection (baseline) and after surgical resection (3 months and 6 months)
  Changes in FEV1 pulmonary function from baseline to 3 and 6 months following lung resection for patients who receive sublobar anatomic resection or are converted to lobectomy.
  FEV1 will be measured using pulmonary function tests and expressed as % of expected value. Changes in FEV1 measured at baseline and at 3 and 6 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ankit Bharat, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No